CLINICAL TRIAL: NCT01885923
Title: Prospective, Randomized, Open, Controlled Study With Information and Telecommunication Technology-aided Relapse Prevention Program in Schizophrenia.
Brief Title: A RCT Study in Schizophrenia Relapse Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prague Psychiatric Center (Other Government)
Responsible Party: Principal Investigator, Filip Spaniel, M.D., Ph.D, MD, Prague Psychiatric Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ITAREPS 2.0; NT/13292 - 3 (Registry Identifier: NT/13292 - 3)
Record Dates: First submitted 2012-08-14; First posted 2013-06-25 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Relapse Schizophrenia
Keywords: schizophrenia; relapse prevention; information technology
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 20% antisychotic dose increase in prodromes (Active Comparator): Antipsychotic dose increase upon prodromes occurence detected by Device- ITAREPS system. All antipsychotics currently registered in Czech Republic will be allowed in this study. All patients will remain on antipsychotic treatment adjusted prior enrollment, so that dose adjustment will be based on their ordinary medication. Participants will be instructed to complete the 10-item EWS Questionnaire upon SMS request sent automatically weekly to their mobile phones. EWSQ detects proportional worsening of the symptoms compared to the last week's score of the questionnaire. Individual EWSQ scores will be sent by participants back to the ITAREPS system as a SMS. If the total score exceeds the given score threshold, an immediate ALERT would be declared and announced to the investigator as an e-mail message and a therapeutic intervention is requested. After detecting the early warning signs by ITAREPS, an immediate 20% increase in the dose of antipsychotic will be required.
  Interventions: Device: ITAREPS
- Treatment as usual (No Intervention): In the control group (treatment-as-usual) participants will not be enrolled in the ITAREPS system.

INTERVENTIONS:
Device: ITAREPS — Program ITAREPS (Information Technology Aided Relaps Prevention in Schizophrenia)
  Other Names: Information Technology Aided Relaps Prevention in Schizophrenia
  Arms: 20% antisychotic dose increase in prodromes

SUMMARY:
THE AIM OF THE PROJECT The main aim lies in the prevention of frequent relapses typical for schizophrenia and schizoaffective disorder by means of simple, highly cost-effective information technology-aided approach RESEARCH HYPOTHESIS A the end of 18 months study duration, patients in the active group enrolled in ITAREPS will demonstrate statistically significantly reduced risk of hospitalization, decreased number of hospitalization days and reduced direct inpatient costs in comparison to control group not using the program.

DETAILED DESCRIPTION:
The ITAREPS 2.0 program employs telecommunication and information technologies in order to detect fluctuations in longitudinal mental health status of patient with schizophrenia and thus signalize the very early stages of prodromes preceding relapse. This approach opens an avenue towards early pharmacological intervention. Subjects (150 patients with diagnosis of schizophrenia and schizoaffective disorder and their family members) will be randomized at a 1:1 ratio into the active or control group. Participants from the active group will be completing two separate versions of the 10-item Early Warning Signs Questionnaire (EWSQ) upon a weekly SMS request generated automatically by the system during 18 months study duration. In this group, automatically generated e-mail alert message feedback to the investigator will be activated in case of prodrome detection, prompting investigator to antipsychotic dose increase by 20%. The control (treatment-as-usual) group will not use ITAREPS system.

ELIGIBILITY:
Inclusion Criteria:

For entry into the study, the following criteria MUST be met:

* Men and women, ages 18 to 60 years, inclusive.
* A diagnosis of schizophrenia or schizoaffective disorder according to ICD-10 classification.
* Having at least TWO psychiatric hospitalization for psychosis before the study enrollment.
* Severity (CGI-S) ≤ 3 at study Visit 1.
* All patients must be on stable doses of antipsychotic medication during the study entry.

Exclusion Criteria:

* Organic mental disorder,
* mental disorder due to psychoactive substance use or mental retardation.
* Participation in another relapse prevention program.
* Hayward compliance rating scale score < 2 at Visit 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective: The hospitalization-free survival rate at 18 months in active group compared to the control group. | 18 months

SECONDARY OUTCOMES:
Number of psychiatric hospitalization days | 18months
Direct impatient costs | 18months
Direct cost of outpatient antipsychotic medication | 18months
Cumulative exposition to antipsychotic medication in both active ITAREPS and control groups | 18months

CONTACTS AND LOCATIONS:
Overall Officials: Filip Spaniel, MD, PhD, Study Director — Prague Psychiatric Center
Locations (1):
- Prague Psychiatric Center, Prague, Czechia

REFERENCES:
- [Derived] Spaniel F, Novak T, Bankovska Motlova L, Capkova J, Slovakova A, Trancik P, Matejka M, Hoschl C. Psychiatrist's adherence: a new factor in relapse prevention of schizophrenia. A randomized controlled study on relapse control through telemedicine system. J Psychiatr Ment Health Nurs. 2015 Dec;22(10):811-20. doi: 10.1111/jpm.12251. Epub 2015 Jul 14. PMID 26176646